CLINICAL TRIAL: NCT03344029
Title: Immunogenicity and Safety of the Shenzhen Trivalent Inactivated Influenza Vaccine Versus a Trivalent Influenza Vaccine Comparator in Healthy Chinese Subjects Aged 18 to 59 Years
Brief Title: Immunogenicity and Safety of the Shenzhen Trivalent Inactivated Influenza Vaccine Versus a Trivalent Influenza Vaccine Comparator in Chinese Subjects 18 to 59 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FST00002; U1111-1183-5912 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Influenza; Flu
Keywords: Influenza; Flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Blind-observer, monocenter, randomized, comparative, Phase IV study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An observer-blind procedure will be followed in the study such that neither the Investigator, subject, nor the Sponsor will know which vaccine has been administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SP Shz TIV (Experimental): Participants aged 18 to 59 years will receive a single injection of SP Shz TIV.
  Interventions: Biological: SP Shz TIV
- Hualan TIV (Active Comparator): Participants aged 18 to 59 years will receive a single injection of Hualan TIV.
  Interventions: Biological: Hualan TIV

INTERVENTIONS:
Biological: SP Shz TIV — 0.5 mL, intramuscular into the deltoid muscle, single injection on Day 0
  Other Names: Sanofi Pasteur Shenzhen Trivalent Influenza Vaccine
  Arms: SP Shz TIV
Biological: Hualan TIV — 0.5 mL, intramuscular into the deltoid muscle, single injection on Day 0
  Other Names: Hualan Trivalent Influenza Vaccine
  Arms: Hualan TIV

SUMMARY:
This was a blind-observer, monocenter, randomized, comparative, Phase IV study designed to evaluate the immunogenicity and safety of the Sanofi Pasteur Shenzhen Trivalent Influenza Vaccine (SP Shz TIV) versus the Trivalent Influenza Vaccine manufactured by Hualan Biological Engineering Inc (Hualan TIV) comparator in healthy Chinese participants aged 18 to 59 years.

DETAILED DESCRIPTION:
This study is designed to demonstrate the non-inferiority of the immune response in terms of geometric mean titers (GMTs) and seroconversion rates for the 3 strains (A/H1N1, A-H3N2, and B) after a single dose of either the SP Shz TIV or Hualan TIV. Vaccine immune responses will be assessed on Day 0 (pre-vaccination) and Day 28 post-vaccination. Solicited reactions will be collected from Day 0 up to Day 7 after vaccination, unsolicited non-serious adverse events (AEs) will be collected from Day 0 up to Day 28 post-vaccination, and serious AEs will be collected from Day 0 up to 6 months post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 to 59 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non- childbearing potential, a female must be post-menopausal for at least 1 year or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine or planned receipt of any vaccine within the period from 2 weeks before trial vaccination to 2 weeks following trial vaccination
* Previous vaccination against influenza (in the previous 6 months) with either the trial vaccines or another vaccine
* Receipt of immune globulins, blood or blood-derived product in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccines components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥ 37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1600 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Summary of Geometric Mean Titers (GMTs) of Each of the Three Strains of TIV Antibodies Following a Single Dose of SP Shz TIV or Hualan TIV | Day 28 post-vaccination
  GMTs were assessed using the hemagglutination inhibition (HAI) assay.
Percentage of Participants with TIV Seroconversion Following a Single Dose of SP Shz TIV or Hualan TIV | Day 28 post-vaccination
  Seroconversion rates were assessed using a HAI assay. Seroconversion was defined as titers <10 (1/dil) at Day 0 and post-injection titer ≥40 (1/dil) at Day 28, or titer ≥10 (1/dil) at Day 0 and a ≥4-fold increase in titer (1/dil) at Day 28.

SECONDARY OUTCOMES:
GMTs of TIV Antibodies Following a Single Dose of SP Shz TIV or Hualan TIV | Day 28 post-vaccination
  GMTs were assessed using the HAI assay.
GMT Ratios of TIV Antibodies Following a Single Dose of SP Shz TIV or Hualan TIV | Day 28 post-vaccination
  GMTs were assessed using the HAI assay.
Percentage of Participants with TIV Antibody Titers ≥10 (1/dil) Following a Single Dose of SP Shz TIV or Hualan TIV | Day 28 post-vaccination
  TIV antibody levels were assessed using the HAI assay.
Percentage of Participants with TIV Antibody Titers ≥40 (1/dil) Following a Single Dose of SP Shz TIV or Hualan TIV | Day 28 post-vaccination
  TIV antibody levels were assessed using the HAI assay.
Percentage of Participants Reporting Solicited Injection site or Systemic Reactions Following a Single Dose of SP Shz TIV or Hualan TIV | Day 0 up to Day 7 post-vaccination
  Solicited injection site reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Shivering

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Sanofi Pasteur Investigational Site 001, Huai'an, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Hu Y, Chu K, Lavis N, Li X, Liang B, Liu S, Shao M, Shu JD, Tabar C, Samson S. Immunogenicity and safety of a trivalent inactivated influenza vaccine produced in Shenzhen, China versus a comparator influenza vaccine: a phase IV randomized study. Hum Vaccin Immunother. 2019;15(5):1066-1069. doi: 10.1080/21645515.2019.1581541. Epub 2019 Apr 2. PMID 30779689